CLINICAL TRIAL: NCT01184872
Title: An Open Label, Multi-center, Randomized, Comparative Phase IIIb Study to Compare Efficacy and Safety of Intravenous (i.v.) Daptomycin With That of Semi-Synthetic Penicillins (SSPs) or Vancomycin in the Treatment of Elderly Patients (Aged ≥ 65 Years) With Complicated Skin and Soft Tissue Infections (cSSTI)
Brief Title: Study to Compare Efficacy and Safety of Daptomycin in Elderly Patients With Complicated Skin and Soft Tissue Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCBC134A2404; 2009-014391-22 (EudraCT Number)
Record Dates: First submitted 2010-02-18; First posted 2010-08-19 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Infections
Keywords: Skin infection; Daptomycin; Elderly; Gram positive; Complicated skin and soft tissue infections
MeSH Terms: conditions — Infections; Cellulitis; Soft Tissue Infections | interventions — Daptomycin; Vancomycin; Oxacillin; Cloxacillin; Floxacillin

ARMS (2):
- Daptomycin (Experimental): Patients with bacteremia: Daptomycin 6 mg/Kg intravenous once daily for at least 5 days and up to 28 days.
  Patients without bacteremia: Daptomycin 4 mg/Kg intravenous once daily for at least 5 days and up to 14 days.
  Interventions: Drug: Daptomycin
- Vancomycin or Semi-Synthetic Penicillins (SSPs) (Active Comparator): Patients with bacteremia: Vancomycin 1 g intravenous twice daily or Semi-Synthetic Penicillins 2 g intravenous every 4 hours for at least 5 days and up to 28 days.
  Patients without bacteremia: Vancomycin 1 g intravenous twice daily or Semi-Synthetic Penicillins 2 g intravenous every 6 hours for at least 5 days and up to 14 days.
  Interventions: Drug: Vancomycin or Semi-Synthetic Penicillins (SSPs)

INTERVENTIONS:
Drug: Daptomycin — Patients with bacteremia: Daptomycin 6 mg/Kg intravenous once daily for at least 5 days and up to 28 days.
  Patients without bacteremia: Daptomycin 4 mg/Kg intravenous once daily for at least 5 days and up to 14 days.
  Arms: Daptomycin
Drug: Vancomycin or Semi-Synthetic Penicillins (SSPs) — Patients with bacteremia: Vancomycin 1 g intravenous twice daily or Semi-Synthetic Penicillins 2 g intravenous every 4 hours for at least 5 days and up to 28 days.
  Patients without bacteremia: Vancomycin 1 g intravenous twice daily or Semi-Synthetic Penicillins 2 g intravenous every 6 hours for at least 5 days and up to 14 days.
  Other Names: Oxacillin,; Cloxacillin,; Flucloxacillin,
  Arms: Vancomycin or Semi-Synthetic Penicillins (SSPs)

SUMMARY:
The purpose of this study is to provide data documenting the efficacy of daptomycin in elderly patients aged ≥ 65 years with complicated Skin and Soft Tissue Infections.

ELIGIBILITY:
Inclusion criteria:

Patients 65 years or older with infection of sufficient severity to require in-patient hospitalization, with parenteral antimicrobial therapy for at least 96 hours.

Patients who have a diagnosis of Gram-positive complicated Skin and Soft Tissue Infections (cSSTIs) with or without bacteremia:

* Wound infections,
* Major abscesses with or without recognized preceding trauma, that require antibiotic therapy in addition to surgical incision and drainage,
* Severe carbunculosis,
* Infected ulcers (except patients with multiple infected ulcers) associated with: diabetes, vascular insufficiency, pressure (i.e., decubitus ulcers).

Exclusion criteria:

Conditions requiring surgery that in and of itself would cure the infection or remove the infected site (e.g., amputation).

Minor or superficial skin infections (e.g., furuncles, simple abscesses, acne, impetigo).

Cellulitis, including erysipelas, not associated with complicating factors. However, patients with cellulitis associated with more serious infection (e.g., surgical wound, diabetic ulcer, deep tissue) can be enrolled (proportion of these patients will be limited to 30%).

Infections for which outcome is difficult to assess:

* Perirectal abscess,
* Hidradenitis suppurativa,
* Gangrene,
* Infected human or animal bites,
* Multiple infected ulcers at distant sites,
* Infected burns (only third degree burn wound or wound area of more than 10 cm diameter),
* Conditions requiring emergency surgery including necrotizing fasciitis.

Medical conditions:

* History of significant allergy or intolerance to Vancomycin or Daptomycin. Hypersensitivity to SSPs penicillins is not an exclusion criterion,
* Concomitant clinically suspected or confirmed other site of infection or disorder at study entry that may interfere with the evaluation in this protocol,
* Infections associated with a permanent prosthetic device that will not be removed within 24 hours after enrolment,
* Known or suspected HIV infection with a CD4+ T-cell count < 500/μL (HIV testing is not required),
* Severe hepatic disease (Child-Pugh Class C) or ALT and/or AST > 5 times ULN and/ or total bilirubin > 2 times ULN at screening,
* Calculated creatinine clearance by the Cockcroft-Gault equation using actual body weight < 30 mL/min or any type of dialysis,
* Treatment with any investigational agent or device within 30 days of study drug administration.

Exclusion criteria related to medications:

* Previous systemic antibacterial therapy for the treatment of Gram-positive complicated skin and soft tissue infections for more than 24 hours within 48 hours prior to the day of first infusion of study drug unless:
* The previous antibacterial therapy was administered for 3 or more calendar days with either worsening or no improvement in the clinical signs and symptoms of cSSTIs, and was not Vancomycin or SSPs.

Other protocol-defined inclusion/exclusion criteria applied.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmceuticals, Study Director — Novartis Pharmceuticals
Locations (17):
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Germany (7):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Pisa, Italy
- Russia (4):
  - Novartis Investigative Site (1), Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site (2), Saint Petersburg
  - Novartis Investigative Site, Yaroslavi
- Spain (3):
  - Novartis Investigative Site (1), Madrid
  - Novartis Investigative Site, Santander
  - Novartis Investigative Site, Seville

REFERENCES:
- [Background] Arbeit RD, Maki D, Tally FP, Campanaro E, Eisenstein BI; Daptomycin 98-01 and 99-01 Investigators. The safety and efficacy of daptomycin for the treatment of complicated skin and skin-structure infections. Clin Infect Dis. 2004 Jun 15;38(12):1673-81. doi: 10.1086/420818. Epub 2004 May 20. PMID 15227611

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daptomycin | Vancomycin or Semi-Synthetic Penicillins (SSPs)
Started | 81 ("Started" indicates randomized and full analysis set.) | 39
Safety Set | 80 (One patient randomized to Daptomycin received Vancomycin.) | 40
Clinical Evaluable Set (CES) | 73 | 30
Microbiologically Evaluable Set (MES) | 65 | 27
Completed | 71 | 31
Not Completed | 10 | 8
Not completed — Adverse Event | 3 | 4
Not completed — Unsatisfactory therapeutic effect | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative problems | 1 | 1
Not completed — Protocol deviation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daptomycin | Vancomycin or Semi-Synthetic Penicillins (SSPs) | Total
Number analyzed (Participants) | 81 | 39 | 120
Age Continuous [Mean (Standard Deviation); unit: years] | 74.63 (6.331) | 75.28 (5.515) | 74.84 (6.063)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 26 | 73
  Male | 34 | 13 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Success at the Test-Of-Cure (TOC) Visit
Description: Success: Clinically significant signs and symptoms associated with the skin infection present at the pre-treatment infection site resolved (cure), or improved without need of further antibacterial therapy. Failure: Persistence or progression of signs and symptoms or development of new clinical signs and symptoms at the infection site, or concomitant antibacterial therapy with activity against isolated organisms, or treatment duration longer than pre-specified, or switch back to intravenous therapy due to relapse, or requirement of a major surgical procedure as adjunct or follow-up therapy.
Time Frame: Baseline and 7 to 14 days after end of therapy
Population: The clinically evaluable population was used for the efficacy analysis. It included all patients who met the criteria for complicated skin and soft tissue, had no substantive protocol deviation, had a sponsor clinical response assessment of "success" or "failure" at the assessment visit, and had a specified baseline primary site of infection.
Measure: Number; unit: participants
Arm/Group | Daptomycin | Vancomycin or Semi-Synthetic Penicillins (SSPs)
Number analyzed (Participants) | 73 | 30
participants
  Success | 65 | 25
  Failure | 8 | 5

2. Secondary Outcome: Number of Participants With Microbiological Response at Test-of-Cure (TOC) Visit
Description: Microbiological Success: All infecting Gram-positive pathogens isolated at baseline were eradicated or presumed to be eradicated at the Test-of-Cure (TOC) evaluation and a super infecting pathogen was not isolated either prior to or at the TOC evaluation. Microbiological Failure: Persistence or relapse / re-infection of one or more infecting Gram-positive pathogens or isolation of a super infecting pathogen prior to or at the TOC evaluation.
Time Frame: Baseline and 7 to 14 days after end of therapy
Population: Population analyzed consisted of patients from the clinically evaluable population who had independent microbiological assessments.
Measure: Number; unit: participants
Arm/Group | Daptomycin | Vancomycin or Semi-Synthetic Penicillins (SSPs)
Number analyzed (Participants) | 65 | 27
participants
  Success | 54 | 23
  Failure | 11 | 4

3. Secondary Outcome: Duration of Treatment (Intravenous)
Description: Duration of treatment is the interval from first to last intravenous (i.v.) administration. It was preferable that a patient complete the whole antibiotic treatment with the randomized i.v. study drug only. Duration of treatment in patients with bacteremia could be extended up to 28 days.
Time Frame: Up to 28 days
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned at randomization.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Daptomycin | Vancomycin or Semi-Synthetic Penicillins (SSPs)
Number analyzed (Participants) | 81 | 39
Days | 7.8 (3.42) | 7.3 (2.42)

4. Secondary Outcome: Duration of Treatment (Intravenous and Oral)
Description: Duration of treatment is the interval from first to last intravenous (i.v.) or to last oral administration if patients switched to an oral antibiotic therapy. It was preferable that a patient complete the whole antibiotic treatment with the randomized i.v. study drug only. Duration of treatment in patients with bacteremia could be extended up to 28 days.
Time Frame: Up to 28 days
Population: The Full Analysis set (FAS) comprised all patients to whom study treatment had been assigned at randomization.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Daptomycin | Vancomycin or Semi-Synthetic Penicillins (SSPs)
Number analyzed (Participants) | 81 | 39
Days
  intravenous only | 7.8 (3.4) | 7.3 (2.4)
  intravenous + oral | 8.7 (4.9) | 9.6 (5.4)

5. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Death
Time Frame: Continuously from baseline up to 28 days after end of antibiotic treatment.
Population: The safety set included all patients who received at least one dose of study medication and who had at least one post-baseline safety assessment.
Measure: Number; unit: participants
Arm/Group | Daptomycin | Vancomycin or Semi-Synthetic Penicillins (SSPs)
Number analyzed (Participants) | 80 | 40
participants
  Adverse Events | 50 | 26
  Serious Adverse Events | 7 | 4
  Death | 0 | 0

ADVERSE EVENTS:
Arm/Group | Daptomycin | Vancomycin or Semi-Synthetic Penicillins (SSPs)
Serious Adverse Events (participants affected / at risk) | 7/80 | 4/40
Other Adverse Events (participants affected / at risk) | 31/80 | 14/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daptomycin (N=80) | Vancomycin or Semi-Synthetic Penicillins (SSPs) (N=40)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Necrosis (General disorders) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Nasopharyngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daptomycin (N=80) | Vancomycin or Semi-Synthetic Penicillins (SSPs) (N=40)
Nausea (Gastrointestinal disorders) | 5 | 2
Hyperthermia (General disorders) | 11 | 3
Blood creatine phosphokinase increased (Investigations) | 5 | 1
Blood creatinine increased (Investigations) | 1 | 2
Blood pressure increased (Investigations) | 5 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypertension (Vascular disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.